CLINICAL TRIAL: NCT02327689
Title: Emtricitabine Plus Adefovir Dipivoxil for Naive Chinese HBV Related Cirrhosis Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Asian-Pacific Alliance of Liver Disease, Beijing (Other)
Collaborators: Beijing Ditan Hospital (Other); Hebei Medical University Pharmaceutical Factory (Industry); National Health and Family Planning Commission, P.R.China (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FTC-01-cirrhosis patients
Record Dates: First submitted 2014-12-23; First posted 2014-12-30 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Hepatitis B, Chronic; Fibrosis
Keywords: Hepatitis B virus; Cirrhosis; Emtricitabine; Adefovir dipivoxil
MeSH Terms: conditions — Hepatitis B, Chronic; Fibrosis; Hepatitis B | interventions — Emtricitabine; adefovir dipivoxil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- compensated HBV related cirrhosis patients (Experimental): Chinese naive compensated HBV related cirrhosis patients were treated with generic emtricitabine capsule(200 mg one time per day) plus adefovir dipivoxil(10 mg one time per day) for 96 weeks
  Interventions: Drug: Emtricitabine plus adefovir dipivoxil
- decompensated HBV related cirrhosis patients (Experimental): Chinese naive decompensated HBV related cirrhosis patients were treated with generic emtricitabine capsule(200 mg one time per day) plus adefovir dipivoxil(10 mg one time per day) for 96 weeks
  Interventions: Drug: Emtricitabine plus adefovir dipivoxil

INTERVENTIONS:
Drug: Emtricitabine plus adefovir dipivoxil — emtricitabine plus adefovir dipivoxil were given to each patients for 96 weeks
  Other Names: Brand name of emtricitabine：Huierding

SUMMARY:
This study evaluates generic emtricitabine(FTC) plus adefovir dipivoxil in Chinese naive HBV related cirrhosis patients. Patients were divided into 2 groups: compensated HBV related cirrhosis patients and decompensated HBV related cirrhosis patients.

DETAILED DESCRIPTION:
Generic emtricitabine(FTC) has been approved for treatment of naive chronic hepatitis B(CHB) patients in China. Yet data are limited for this agent plus adefovir dipivoxil in cirrhosis patients. The investigators design this trial to test the effect of FTC plus adefovir dipivoxil in Chinese naive compensated and decompensated HBV related cirrhosis patients.

ELIGIBILITY:
Inclusion Criteria:

* Dignosed cirrhosis patients
* HBsAg positive for more than 6 months
* HBV DNA detectable
* Nucleoside/nucleotide naive patients

Exclusion Criteria:

* Diagnosed HCC with AFP and ultrasound, CT or MRI
* Creatine >130μmol/L or Ccr < 70mL/min
* Hemoglobin <100g/L
* Coinfected with HAV,HEV,HCV,HDV or HIV
* ANA > 1:100
* Uncontrolled cardiovascular diseases, kidney diseases,lung diseases, neurological diseases, digestive diseases,metabolic disorders, immune-compromised diseases or cancer;
* Drug abuse or alcohol addiction
* Previous history of taking agents of lamivudine, adefovir, tenofovir entecavir or telbivudine
* Long-term use of immunosuppressor or immunomodulator 6 months before enrollment to this trial
* Underwent liver transplantation or liver transplantation in schedule
* Allergic to nucleoside or nucleotide analogues
* Pregnancy or in breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
virological response rate | week 96
  HBV DNA < 500 copies/ml

SECONDARY OUTCOMES:
HBV DNA negativity rate | week 24, 48 and 72
  HBV DNA < 500 copies/ml
HBV DNA decrease level | week24, 48, 72 and 96
  HBV DNA decrease compared with baseline（log10 copies/ml）
biochemical response | week 24,48,72 and 96
  ALT normalization
HBeAg loss | week 24,48,72 and 96
  HBeAg loss in HBeAg positive group
HBeAg seroconversion | week 24,48,72 and 96
  HBeAg seroconversion in HBeAg positive group
HBeAg reversion | week 24,48,72 and 96
  HBeAg positive in Baseline HBeAg negativie group patients
HBsAg loss | week 24,48,72 and 96
  HBsAg loss in both group
HBsAg seroconversion | week 24,48,72 and 96
  HBsAg loss and anti-HBs positive
HBV genetic resistance to emtricitabine and adefovir | week 24,48,72 and 96
  HBV genetic resistance to emtricitabine and adefovir
adverse event | week 24,48,72 and 96
  type and rate of adverse events;type and rate of severe adverse event
incidence of HCC | week 24,48,72 and 96
  incidence of HCC in both groups
change of MELD score and Child-Pugh score | week 24,48,72 and 96
  change of MELD score and Child-Pugh score in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Jun Cheng, M.D., Principal Investigator — Asian Pacific Alliance of Liver Diseases, Beijing

REFERENCES:
- [Background] Gish RG, Leung NW, Wright TL, Trinh H, Lang W, Kessler HA, Fang L, Wang LH, Delehanty J, Rigney A, Mondou E, Snow A, Rousseau F. Dose range study of pharmacokinetics, safety, and preliminary antiviral activity of emtricitabine in adults with hepatitis B virus infection. Antimicrob Agents Chemother. 2002 Jun;46(6):1734-40. doi: 10.1128/AAC.46.6.1734-1740.2002. PMID 12019083
- [Background] Lim SG, Ng TM, Kung N, Krastev Z, Volfova M, Husa P, Lee SS, Chan S, Shiffman ML, Washington MK, Rigney A, Anderson J, Mondou E, Snow A, Sorbel J, Guan R, Rousseau F; Emtricitabine FTCB-301 Study Group. A double-blind placebo-controlled study of emtricitabine in chronic hepatitis B. Arch Intern Med. 2006 Jan 9;166(1):49-56. doi: 10.1001/archinte.166.1.49. PMID 16401810